CLINICAL TRIAL: NCT00448058
Title: A Ten-Week, Multicenter, Randomized, Double-Blind, Placebo and Active-Controlled, Parallel-Group, Flexible-Dose Study Evaluating the Efficacy, Safety, and Tolerability of GSK372475 (1.5 mg/Day to 2.0 mg/Day) or Extended Release Venlafaxine XR (150 mg/Day to 225 mg/Day) Compared to Placebo in Adult s
Brief Title: A Study Of New Medicine (GSK 372475) For The Treatment Of Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SND 103285
Record Dates: First submitted 2007-03-13; First posted 2007-03-15 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2011-11

CONDITIONS: Depressive Disorder
Keywords: Flexible-dose; GSK372475; MDD; Venlafaxine XR; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major | interventions — GSK372475; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- GSK372475 (Experimental): flexible-dose design from GSK372475 1.0 mg/day to GSK372475 2.0 mg/day
  Interventions: Drug: GSK372475
- Venlafaxine (Active Comparator): Flexible- dose design from Venlafaxine XR 75 mg/day to Venlafaxine XR 225 mg/day
  Interventions: Drug: venlafaxine
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GSK372475 — daily administration during the 10-week treatment phase
  Arms: GSK372475
Drug: venlafaxine — daily administration during the 10-week treatment phase
  Arms: Venlafaxine
Drug: placebo — daily administration during the 10-week treatment phase
  Arms: placebo

SUMMARY:
To evaluate the efficacy, safety, and tolerability of GSK372475 compared with placebo in the treatment of outpatient subjects with Major Depressive Disorder (MDD)

DETAILED DESCRIPTION:
A Ten-Week, Multicenter, Randomized, Double-Blind, Placebo and Active-Controlled, Parallel-Group, Flexible-Dose Study Evaluating the Efficacy, Safety, and Tolerability of GSK372475 (1.5 mg/day to 2.0 mg/day) or Extended Release Venlafaxine XR (150 mg/day to 225 mg/day) Compared to Placebo in Adult Subjects Diagnosed with Major Depressive Disorder

ELIGIBILITY:
Inclusion Criteria:

* Major depressive episode (MDE) associated with Major Depressive Disorder (DSM-IV-TR criteria)
* Duration of current episode is at least 12 weeks duration and less than 2 years
* Symptoms of decreased energy, pleasure, and interest
* Female subjects who agree to use acceptable methods of birth control throughout the study

Exclusion criteria:

* Current diagnosis of Panic Disorder, or symptoms of generalized anxiety or panic attacks that could interfere with their ability to complete the trial
* Symptoms of MDE better accounted for by another diagnosis
* Diagnosis of Bipolar, schizophrenia, other psychotic disorder(s), borderline or antisocial personality disorder, or dementia.
* Started psychotherapy within 3 months prior to the Screening
* Received electroconvulsive therapy or transcranial magnetic stimulation within 6 months prior to screening
* Received psychoactive drugs within 4 weeks of randomization
* Positive urine drug screen or positive blood alcohol
* Suicidal risk or has had any previous suicide attempt, a family history of suicide attempt
* Positive pregnancy test
* History of seizure disorder, myocardial infarction (< 1yr), or unstable medical condition
* Failed to respond to an adequate course of pharmacotherapy of at least 2 different antidepressants

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 396 (Actual)
Dates: Start 2007-04; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Change from randomization to the end of the Treatment Phase (Week 10) on a depression rating scale. | Randomisation (week 0) And end of the treatment

SECONDARY OUTCOMES:
Endpoints related to response & remission on depression rating scales during time of treatment exposureChange during treatment & at endpoint-week 10:in Clinical Global Impression scale; in motivation, energy, & sexual functioning on patient-rated scales | Randomisation (week 0) and at weeks 1,2,4,6,8 and week 10 (end of treatment phase)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (40):
- Australia (4):
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Kippa-Ring, Queensland
  - GSK Investigational Site, Epping, Victoria
  - GSK Investigational Site, Heidelberg West, Victoria
- Belgium (2):
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Mont-Godinne
- Bulgaria (2):
  - GSK Investigational Site, Burgas
  - GSK Investigational Site, Varna
- Canada (6):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Sydney, Nova Scotia
  - GSK Investigational Site, Burlington, Ontario
  - GSK Investigational Site, Mississauga, Ontario
  - GSK Investigational Site, Montreal, Quebec
- Estonia (3):
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
  - GSK Investigational Site, Võru
- Finland (2):
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Turku
- France (3):
  - GSK Investigational Site, Arcachon
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Toulouse
- Germany (5):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Unterhaching, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Westerstede, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
- India (4):
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Chennai
  - GSK Investigational Site, Hyderabad
  - GSK Investigational Site, Tirupati
- Poland (4):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Skorzewo
- Slovakia (2):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Michalovce
- South Africa (3):
  - GSK Investigational Site, Observatory ,Cape Town
  - GSK Investigational Site, Somerset West
  - GSK Investigational Site, Vereeniging

REFERENCES:
- [Background] Learned S, Graff O, Roychowdhury S, Moate R, Krishnan KR, Archer G, Modell J, Alexander R, Zamuner S, Lavergne A, Evoniuk G, Ratti E. Results of Two Double-Blind, Placebo- and Active-Controlled Studies of GSK372475, a Triple Monoamine Reuptake Inhibitor, in the Treatment of Major Depressive Disorder. [J Psychopharmacol EPublication ahead of print. DOI 10.1177/0269881111424931]. 2011;
- [Derived] Learned S, Graff O, Roychowdhury S, Moate R, Krishnan KR, Archer G, Modell JG, Alexander R, Zamuner S, Lavergne A, Evoniuk G, Ratti E. Efficacy, safety, and tolerability of a triple reuptake inhibitor GSK372475 in the treatment of patients with major depressive disorder: two randomized, placebo- and active-controlled clinical trials. J Psychopharmacol. 2012 May;26(5):653-62. doi: 10.1177/0269881111424931. Epub 2011 Nov 2. PMID 22048884